CLINICAL TRIAL: NCT03384758
Title: Evaluation of the Effect of Compression Therapy on the Microcirculation in Patients With Leg Edema and Mild to Moderate PAD or Diabetes Mellitus.
Brief Title: Evaluation of Compression Therapy in Patients With Mild to Moderate PAD or Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Erlangen (Other)
Responsible Party: Principal Investigator, Ulrich Rother, Principal investigator PD Dr. med. Ulrich Rother, University Hospital Erlangen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Perfusion under Compression
Record Dates: First submitted 2017-12-12; First posted 2017-12-27 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Peripheral Arterial Disease; Diabetes Mellitus; Leg Edema
Keywords: Compression therapy; Microcirculation; Diabetes mellitus; Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease; Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- mild to moderate PAD (Active Comparator)
  Interventions: Device: Compression Therapy
- Diabetes mellitus (Active Comparator)
  Interventions: Device: Compression Therapy
- Healthy volunteers (Placebo Comparator)
  Interventions: Device: Compression Therapy

INTERVENTIONS:
Device: Compression Therapy — Therapy of the leg edema with compression stockings class I for three hours, after a short break with compression stocking class II for again three hours.

SUMMARY:
Aim of this prospective clinical study is the Evaluation of the Effect of Compression Therapy on the Microcirculation in Patients With Leg Edema and Mild to Moderate PAD or Diabetes Mellitus.

DETAILED DESCRIPTION:
Aim of this prospective clinical study is the Evaluation of the Effect of Compression Therapy on the Microcirculation in Patients With Leg Edema and Mild to Moderate PAD or Diabetes Mellitus. The microcirculation should be assessed by a combination of laserdoppler flowmetry and white light tissue spectrometry (O2C Device, Parameters sO2, Flow, rHb). By this, it is possible to detect the influence of the compression therapy on the skin microcirculation.

Therefore, three study arms should be investigated, all patients clinically suffering under leg edema: healthy volunteers, patients with mild to moderate PAD and diabetics. All patients are recieveing compression therapy (Compression stockings class I for three hours, after a short break compression stockings class II for 3 hours) under Perfusion assessment control (O2C device).

ELIGIBILITY:
Inclusion Criteria:

Study-Arm PAD:

* leg edema
* symptomatic PAD (Fontaine stage II)
* no palpable foot pulses
* ABI <0.9 and >0.6, absolute ankle pressure > 60mmHg

Study-Arm Diabetes:

* leg edema
* Diabetes mellitus Typ 2 (history of longer than 2 years)
* palpable foot pulses
* Pallaesthesie >6
* Wagner Score 0

Exclusion Criteria:

Study-Arm PAD:

* Critical limb ischemia
* ABI < 0.6
* simoultaneous Diabetes Mellitus

Study-Arm Diabetes:

* Wagner Score >0
* Pallasthesie <6

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by questionnaire | 12 Months
  The Adverse Events are defined in the questionnaire as: Abort of the Therapy, Pressure marks, Quantification of the wearing comfort (Points 1-10), subjective reduction of the leg edema (Points 1-10)
sO2 | 12 Months
  The Perfusion Situation should be recorded on the Level of Microcirculation by the Parameter sO2
Flow | 12 Months
  The Perfusion Situation should be recorded on the Level of Microcirculation by the Parameter Flow
rHb | 12 Months
  The Perfusion Situation should be recorded on the Level of Microcirculation by the Parameter rHb

CONTACTS AND LOCATIONS:
Locations (1):
- University of Erlangen, Vascular Surgery, Erlangen, Germany

REFERENCES:
- [Derived] Rother U, Grussler A, Griesbach C, Almasi-Sperling V, Lang W, Meyer A. Safety of medical compression stockings in patients with diabetes mellitus or peripheral arterial disease. BMJ Open Diabetes Res Care. 2020 Jun;8(1):e001316. doi: 10.1136/bmjdrc-2020-001316. PMID 32503811